CLINICAL TRIAL: NCT02694497
Title: Understanding Transmission of Genital and Extra-genital Chlamydia Trachomatis Infections in Women Receiving Routine Care; Implications for Control Strategies
Brief Title: Transmission of Genital and Extra-genital Chlamydia Trachomatis Infections in Women
Acronym: FemCure
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Public Health Service South Limburg (Other Government); Public Health Service Rotterdam (Unknown); Public Health Service of Amsterdam (Other Government); National Institute for Public Health and the Environment (RIVM) (Other Government); STIAIDSNetherlands (Unknown)
Responsible Party: Sponsor
Other Study IDs: FemCure
Record Dates: First submitted 2016-02-15; First posted 2016-02-29 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2017-08

CONDITIONS: Chlamydia Trachomatis Infection
Keywords: transmission; women; genital; anorectal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will collect a self-administered anorectal and vaginal swab at 8 time-points: pre-treatment during the visit at the STI clinic at which the treatment is given (T0), and at the end of weeks 1, 2, 4, 6, 8, 10, and 12. At T0, T4, T8 and T12 (visits at the clinic), the participants take an additional self-administered anorectal and vaginal swab that is otherwise exactly the same as the home-taken samples, but stored in a different buffer and processed immediately, i.e. cooled at -80°C within 24 hours, to allow CT viability testing. At the clinic visit, we will also consider to obtain a nurse-taken pharyngeal swab for later CT testing. For self-collection of the anorectal and genital samples, participants receive clear instructions.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Chlamydia care as usual

SUMMARY:
Multicenter prospective cohort study in Chlamydia trachomatis positive women after regular treatment to understand the transmission of anorectal CT infections.

DETAILED DESCRIPTION:
Rationale:

Current national and international strategies for the control of Chlamydia trachomatis (CT) critically fail to obtain a reduction in transmission. In women, anorectal infections are about as common as genital CT. Yet anorectal CT remain untested as sexually transmitted infection (STI) clinics, general practitioners, hospital and population testing initiatives largely focus on genital CT. Part of untested anorectal CT is incidentally treated with the treatments applied for genital CT, as in women anorectal CT is often concurrent with genital CT. Yet, it is unknown whether transmission of anorectal CT can still occur after currently recommended treatment. Anorectal and genital CT were observed quite often after regular treatment (up to 40% detection by nucleic acid amplification tests-NAAT). Proposed reasons for such detection include a new (re-)infection from a partner or self-infection from another anatomic, e.g. anorectal, site. Anorectal infections are a potential reservoir for ongoing transmission of genital and anorectal CT in the population, between partners and between anatomic sites of an individual. Yet, neither the transmission potential nor the transmission impact of anorectal infections has been reported. The scientific evidence for the optimal control strategy for anorectal CT and thereby CT in its totality, is lacking.

Objective:

To understand the transmission of anorectal CT infections in women, i.e. from their male sexual partner(s) and from and to the genital region of the same woman, in women who receive routine care, in order to inform guidelines to optimize CT control.

Study population:

Participants are recruited from 3 large Dutch STI clinics, in South Limburg, Amsterdam and Rotterdam. Eligible participants are likely to reflect the STI clinic population, in terms of age, ethnicity and level of education. Participants include genital and/or anorectal CT positive women (n=400).

Study design:

A multicentre prospective cohort study is set up with biological and behavioural measurements after routine treatment of CT. During 3 months, the participants will be studied using a self-administered anorectal and vaginal swab that is self-collected pre-treatment (T0), and at the end of weeks 1, 2, 4, 6, 8, 10, and 12. Samples are tested using NAAT for presence of CT-DNA (detection), concentration (load), viability (weeks 4,8, and 12), and CT type (multilocus sequence typing-MLST) to confirm re-infection. To validate sexual exposure, chromosomal Y DNA (as a marker for semen exposure) in genital and anorectal samples is applied. At each sampling time, online self-administered questionnaires on behaviour (e.g. anorectal exposure) and symptoms will be completed.

Outcomes:

The outcome is detection of anorectal and genital CT at any of the time -points.

Primary outcome is incident detection by NAAT, and secondary outcomes include detection of viable CT and CT-DNA concentration.

Statistical analyses:

In statistical analyses, using logistic regression models, the impact of two key factors will be assessed (i.e. sexual exposure and alternate anatomic site of infection) on detection of anorectal and genital CT. In sub-analyses, the role of treatment-type is evaluated.

Expected results:

This project will provide scientific insight in the role of anorectal CT in maintaining the CT burden, and it will provide practical recommendations (STI guidelines) to reduce avoidable transmission. Implications will be to improve care strategies for (re-)testing and partner management that currently largely neglect anorectal CT, benefitting the individual (better fitting care) and public health (reducing burden) and eventually cost-effectiveness of care.

ELIGIBILITY:
Inclusion Criteria:

* Chlamydia trachomatis test positive (genital and or anorectal)

Exclusion Criteria:

* (reported) co-infection with gonorrhoea
* (reported) co-infection with HIV
* (reported) co-infection with syphilis
* (reported) pregnant
* (reported) anti-Chlamydial antibiotic use (period screening-treatment)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are recruited from 3 large Dutch STI clinics, in South Limburg, Amsterdam and Rotterdam. Eligible participants are likely to reflect the STI clinic population, in terms of age, ethnicity and level of education. Participants include genital and/or anorectal CT positive women (n=400).
Sampling Method: Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Detection of Chlamydia after treatment. | 0-12 weeks after regular treatment
  Detection of anorectal and genital CT by NAAT

SECONDARY OUTCOMES:
Culture of Chlamydia after treatment | 0-12 weeks after regular treatment
  Detection of viable CT
Viability PCR of Chlamydia after treatment | 0-12 weeks after regular treatment
  Detection of viable CT
CT concentration after treatment | 0-12 weeks after regular treatment
  CT-DNA concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Service South Limburg, Geleen, South Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Not yet

REFERENCES:
- [Result] Dukers-Muijrers NH, Wolffs PF, Eppings L, Gotz HM, Bruisten SM, Schim van der Loeff MF, Janssen K, Lucchesi M, Heijman T, van Benthem BH, van Bergen JE, Morre SA, Herbergs J, Kok G, Steenbakkers M, Hogewoning AA, de Vries HJ, Hoebe CJ. Design of the FemCure study: prospective multicentre study on the transmission of genital and extra-genital Chlamydia trachomatis infections in women receiving routine care. BMC Infect Dis. 2016 Aug 8;16:381. doi: 10.1186/s12879-016-1721-x. PMID 27502928
- [Derived] Janssen KJH, Wolffs PFG, Hoebe CJPA, Heijman T, Gotz HM, Bruisten SM, Schim van der Loeff M, de Vries HJ, Dukers-Muijrers NHTM. Determinants associated with viable genital or rectal Chlamydia trachomatis bacterial load (FemCure). Sex Transm Infect. 2022 Feb;98(1):17-22. doi: 10.1136/sextrans-2020-054533. Epub 2021 Jan 13. PMID 33441449
- [Derived] Dukers-Muijrers NHTM, Wolffs P, Lucchesi M, Gotz HM, De Vries H, Schim van der Loeff M, Bruisten SM, Hoebe CJPA. Oropharyngeal Chlamydia trachomatis in women; spontaneous clearance and cure after treatment (FemCure). Sex Transm Infect. 2021 Mar;97(2):147-151. doi: 10.1136/sextrans-2020-054558. Epub 2020 Jul 31. PMID 32737209
- [Derived] Dukers-Muijrers NHTM, Janssen KJH, Hoebe CJPA, Gotz HM, Schim van der Loeff MF, de Vries HJC, Bruisten SM, Wolffs PFG. Spontaneous clearance of Chlamydia trachomatis accounting for bacterial viability in vaginally or rectally infected women (FemCure). Sex Transm Infect. 2020 Nov;96(7):541-548. doi: 10.1136/sextrans-2019-054267. Epub 2020 Feb 17. PMID 32066588
- [Derived] Dukers-Muijrers NHTM, Wolffs PFG, de Vries HJC, Gotz HM, Janssen K, Hoebe CJPA. Viable Bacterial Load Is Key to Azithromycin Treatment Failure in Rectally Chlamydia trachomatis Infected Women (FemCure). J Infect Dis. 2019 Sep 13;220(8):1389-1390. doi: 10.1093/infdis/jiz267. No abstract available. PMID 31107956
- [Derived] Dukers-Muijrers NHTM, Wolffs PFG, De Vries H, Gotz HM, Heijman T, Bruisten S, Eppings L, Hogewoning A, Steenbakkers M, Lucchesi M, Schim van der Loeff MF, Hoebe CJPA. Treatment Effectiveness of Azithromycin and Doxycycline in Uncomplicated Rectal and Vaginal Chlamydia trachomatis Infections in Women: A Multicenter Observational Study (FemCure). Clin Infect Dis. 2019 Nov 13;69(11):1946-1954. doi: 10.1093/cid/ciz050. PMID 30689759
- See also: published study design — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4977887/pdf/12879_2016_Article_1721.pdf